CLINICAL TRIAL: NCT06709612
Title: Pilot Phase II Study of AMT-143 for Postsurgical Analgesia After Hernia Repair
Brief Title: Postsurgical Analgesia After Hernia Repair
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: AmacaThera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AMT-143-002
Record Dates: First submitted 2024-10-31; First posted 2024-11-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hernia Repair; Hernia Inguinal; Hernia Surgery; Hernia, Inguinal/Surgery; Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal; Hernia | interventions — Sodium Chloride; Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AMT-143 (Experimental)
  Interventions: Drug: AMT-143
- Saline Placebo (Placebo Comparator)
  Interventions: Other: Saline (NaCl 0,9 %) (placebo)
- Ropivacaine solution (Active Comparator)
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: AMT-143 — AMT-143 is provided as a hydrogel containing 385 mg/mL ropivacaine (on a ropivacaine hydrochloride equivalence basis).
  Participants undergoing primary open hernia repair, will be randomized to one of three treatment cohorts of escalating doses of AMT-143 hydrogel:
  * Cohort 1: 1 mL AMT-143 hydrogel
  * Cohort 2: 2 mL AMT-143 hydrogel
  * Cohort 3: 3 mL AMT-143 hydrogel
  Arms: AMT-143
Other: Saline (NaCl 0,9 %) (placebo) — Saline placebo will consist of 0.9% sodium chloride injection USP and will be administered in an amount matching the volume of AMT-143 to be used in each of the Cohorts 1 to 3.
  Arms: Saline Placebo
Drug: ropivacaine — The active comparator, ropivacaine hydrochloride 1% solution will be administered at a volume of 5 mL (50 mg) for all 3 cohorts.
  Arms: Ropivacaine solution

SUMMARY:
The study is designed to evaluate the safety, efficacy, and pharmacokinetics (PK) of three ascending doses of AMT-143 to determine the appropriate dose of AMT-143 for the management of postsurgical pain following inguinal hernia repair.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria apply to all participants scheduled for open inguinal hernia repair in all cohorts.

1. Provides voluntary written informed consent.
2. Participants are ≥18 years of age at screening.
3. Scheduled to undergo unilateral open inguinal hernia repair.
4. Body mass index (BMI) ≤40.0 kg/m2.
5. Male participants must be sterile (biologically or surgically) or commit to the use of a reliable method of birth control for the duration of the study until at least 1 week after the administration of study medication.
6. Female participants:

   * Not pregnant (female participant of childbearing potential must have a negative urine pregnancy test before surgery).
   * Not lactating.
   * Not planning to become pregnant during the study.
   * Be surgically sterile; or at least two years post-menopausal; or have a monogamous partner who is surgically sterile; or is practicing double-barrier contraception; or practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity); or using an insertable, injectable, transdermal, or combination oral contraceptive approved by Health Canada for greater than 2 months prior to screening visits and commits to the use of an acceptable form of birth control for the duration of the study.
7. In the opinion of the Investigator, is willing and able to understand the study procedures, and agrees to adhere to the requirements of the study protocol, in order to enable accurate and appropriate responses to pain scales.

Exclusion Criteria:

The following exclusion criteria apply to all participants in all cohorts.

1. Have chronic pain and have been receiving or have received chronic opioid therapy defined as greater than 15 morphine equivalents units per day for greater than 3 out of 7 days per week over a one-month period within 12 months of study treatment initiation.
2. History of hypersensitivity to any ingredient in the formulation (hyaluronan or methylcellulose).
3. History of hypersensitivity or allergy to amide type local anaesthetics (lidocaine, bupivacaine, or ropivacaine).
4. History of ventricular tachycardia, ventricular fibrillation, or atrioventricular block without a pacemaker.
5. Have a clinically significant abnormal clinical laboratory test value, according to the judgement of the investigator.
6. Have a clinically significant 12-lead ECG abnormality, according to the judgement of the investigator.
7. Have received any medications with a potential for drug interactions with ropivacaine (i.e., amide-type local anaesthetics such as lidocaine, bupivacaine, mepivacaine and prilocaine; antiarrhythmics such as procainamide, disopyramide, tocainide, mexiletine and flecainide; sedative; strong inhibitors of cytochrome P4501A2 such as fluvoxamine enoxacin, theophylline and imipramine for at least 5 half-lives prior to the start of this).
8. Have received any investigational product within 30 days before dosing with study medication.
9. Suspected or known history of substance abuse and/or alcoholism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-27 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events to evaluate the safety and tolerability of AMT-143 | From surgery to Day 28 follow-up
  To evaluate the safety and tolerability of AMT-143 for postsurgical pain management following inguinal hernia repair surgery.
  The safety endpoint of the study will be the incidence of Treatment Emergent Adverse Events (TEAEs). This will include reported Adverse Events as well as all clinically significant abnormalities in clinical laboratory investigations, vital signs, physical examination results, and ECG tracings.
Pharmacokinetics of AMT-143 | From surgery to Day 28 follow-up
  To assess the PK profile of AMT-143. Plasma samples will be analyzed for ropivacaine concentrations using a validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) method. Incurred sample reanalysis will be performed on approximately 10% of study samples with a minimum of 20 samples for confirmation of results. At least two thirds of the incurred samples analyzed should have a percent difference between re-assay & original concentrations within ±20%. Plasma concentration-time data for AMT-143 will be analyzed by the noncompartmental method to obtain the PK parameters using validated Phoenix WinNonlin® version 8.3 or higher software (Pharsight Corp).

SECONDARY OUTCOMES:
Analgesic efficacy of AMT-143 | From surgery to Day 28 follow-up
  To evaluate analgesic efficacy of AMT-143 for postsurgical pain management following inguinal hernia repair surgery utilizing the Numeric Rating Scale (NRS).
  The NRS runs from 0 (no pain) to 10 (worst pain).

IPD SHARING:
Plan to Share IPD: No
Pilot study with limited enrollment.